CLINICAL TRIAL: NCT06051123
Title: Effects of Probiotics on Lipidomic Profile and Disease Evolution in ALS-FTDSD Patients: A Randomized Multicenter, Double-blind, Phase II, Placebo-controlled, Parallel Trial.
Brief Title: Effects of Probiotics in Amyotrophic Lateral Sclerosis-Frontotemporal Dementia Spectrum Disorder (ALS-FTDSD) Patients
Acronym: PROBIOTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2024-11453
Record Dates: First submitted 2023-08-11; First posted 2023-09-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: ALSFTD
Keywords: ALS; FTD; motor function; probiotics; lipidomics; metabolites; neurofilament; microbiome
MeSH Terms: conditions — Frontotemporal Dementia With Motor Neuron Disease | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Phase 2 study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this group will be randomized to receive a probiotic formulation for 24 weeks.
  Interventions: Dietary Supplement: Probiotic
- Control Group (Placebo Comparator): Participants in this group will be randomized to receive a placebo for 24 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants will be taking 1 sachet a day.
  Arms: Experimental Group
Dietary Supplement: Placebo — Participants will be taking 1 sachet a day.
  Arms: Control Group

SUMMARY:
The aim of this study is to assess the impact of a probiotic formulation on participants with ALS-FTDSD. It is hypothesized that participants given the probiotics will have different lipid profiles compared to participants receiving the placebo at different time points.

DETAILED DESCRIPTION:
Individuals with ALS-FTDSD and healthy individuals can participate in this randomized, double-blind, parallel, placebo-controlled study. Participants will be enrolled for a period of 32 weeks, with an intervention period of 24 weeks. For ALS-FTDSD participants, there will be 9 visits during the intervention (5 in-person and 4 phone calls) and 1 follow-up call post-intervention. For healthy participants, there will be 4 in-person visits. For all participants, in-person visits will involve filling out questionnaires, giving blood samples, and returning stool samples.

ELIGIBILITY:
Inclusion Criteria:

ALS participants:

1. Aged 18 years old or greater.
2. Diagnosis of ALS by El Escorial Criteria revised (possible, probable, probable with lab support and definite).
3. Onset of weakness or speech impairment no more than 24 months before randomization.
4. ALSFRS-R equal or superior to 24/48 at screening, with no more than one subscore under 2/4. ALSFRS-R slope of decline of at least 0.5 points per month on the ALSFRS- R, calculated as (48-score at screening)/ (months since onset of weakness).
5. SVC greater than or equal to 60% predicted for sex, age and height at screening.
6. Note on FTD Symptoms: The presence of FTD symptoms is not a requirement for inclusion in this study. Participants with a diagnosis of ALS, whether or not accompanied by FTD symptoms, are eligible for inclusion. No prior or screening diagnosis of FTDSD is required.
7. Subject has an informant/caregiver who has frequent and sufficient contact to provide accurate information about the patient's cognitive abilities and behaviors to complete the ALS-CBS.
8. Participants apt to comprehend and sign the ICF.
9. Participants of child-bearing potential must have a negative urine pregnancy test at screening and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

   1. Abstinence or agrees to use contraception if planning to become sexually active.
   2. Hormonal contraceptives including oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormone implant
   3. Double-barrier method
   4. Intrauterine devices
   5. Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   6. Vasectomy of partner at least 6 months prior to screening
10. Willing to maintain eating habits throughout the study.
11. Willing to refrain from consuming probiotic supplements and food containing added probiotics and/or prebiotics (e.g., yogurts with live, active cultures or supplements) from the moment of screening until the end of the study.

Healthy controls:

1. Aged 18 years old or greater.
2. Able to comprehend and willing to sign ICF.
3. Participants of child-bearing potential must have a negative urine pregnancy test at screening and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

   1. Abstinence or agrees to use contraception if planning to become sexually active.
   2. Hormonal contraceptives including oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormone implant
   3. Double-barrier method
   4. Intrauterine devices
   5. Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   6. Vasectomy of partner at least 6 months prior to screening
4. Willing to maintain eating habits throughout the study.
5. Willing to refrain from consuming probiotic supplements and food containing added probiotics and/or prebiotics (e.g., yogurts with live, active cultures or supplements) from the moment of screening until the end of the study

Informants/caregivers:

1. Aged 18 years old or greater.
2. Has frequent and sufficient contact to provide accurate information about the patient's cognitive abilities and behaviors to complete the ALS-CBS.
3. Able to comprehend and willing to sign ICF.

Exclusion Criteria:

ALS Participants:

1. Use of respiratory support (non-invasive ventilation or mechanical respiratory support) at screening.
2. Significant medical condition or behavioral issues that could interfere with participation in the clinical trial in the principal investigator's opinion.
3. Use of a feeding tube at randomization.
4. Use of lipid-lowering drugs for less than 3 months before randomization.
5. Introduction of lipid-lowering drug unless it is due to the event of acute coronary syndrome or stroke as per Canadian guidelines.
6. Use of edaravone with stable dosage for less than 2 months before randomization.
7. Use of riluzole, or ALBRIOZA™ with stable dosage for less than 1 month before randomization.
8. Introduction of edaravone, riluzole or ALBRIOZA™ during the clinical trial.
9. Immunodeficiency (immune-compromised and immune-suppressed participants, e.g., AIDS, lymphoma, participants undergoing long-term corticosteroid treatment, chemotherapy and allograft participants).
10. Pregnancy (as per serum HCG pregnancy test at screening), planning to be pregnant or currently breastfeeding.
11. Use of probiotics other than the study medication in the month prior to randomization.

    Note: participants could be eligible to participate after a 4-week washout period.
12. Use of any antibiotic drug in the month prior to randomization. Note: participants could be eligible to participate after a 4-week washout period.
13. Milk and soy allergy, or severe lactose intolerance.
14. Currently enrolled in another clinical trial.

Healthy Participants:

1. Use of lipid-lowering drugs for less than 3 months before randomization.
2. Introduction of lipid-lowering drug unless it is due to the event of acute coronary syndrome or stroke as per Canadian guidelines.
3. Pregnancy (as per serum HCG pregnancy test at screening), planning to be pregnant or currently breastfeeding. Note: participants will not take the IP or placebo, but pregnancy is a major factor that could affect lipidomic profiling.
4. Use of probiotics in the month prior to day 0 of the study (visit 2). Note: participants could be eligible to participate after a 4-week washout period. Although participants will not consume any study product, we aim to maintain environmental factors comparable to the ALS-FTDSD group.
5. Use of any antibiotic drug in the month prior to day 0 of the study (visit 2). Note:

   participants could be eligible to participate after a 4-week washout period. Although participants will not consume any study product, we aim to maintain environmental factors comparable to the ALS-FTDSD group.
6. Milk and soy allergy, or severe lactose intolerance. Note: Although participants will not consume any study product, we aim to maintain environmental factors comparable to the ALS-FTDSD group. We aim to exclude allergies, so participants are maintained on standard diet.
7. Currently enrolled in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in lipidomic profiles | 24 weeks
  To compare the change in lipidomic profiles from baseline in the probiotic and placebo groups (within-group) as well as in between-group differences over the 24 weeks of intervention. This will be a lipid profiling and quantification by using mass-spectrometry-based lipidomics. We are going to test 900 different lipids, which can be classified in 20 classes ans subclasses of interest.
Change in polar metabolite profiles | 24 weeks
  To compare the change in polar metabolite profiles from baseline in the probiotic and placebo groups (within-group) as well as in between-group differences over the 24 weeks of intervention. Targets will be key microbiota metabolites: trimethylamine N-oxide (TMAO), short-chain fatty acids, and metabolites derived from tryptophan.

SECONDARY OUTCOMES:
Change in ALSFRS-R score | 24 weeks
  To compare the average change from baseline in the rate of decline in ALS Functional Rating Scale Revised (ALSFRS-R) between the probiotic and placebo groups over the 24 weeks of intervention.
Change in ALS-CBS score | 24 weeks
  To compare the average change from baseline in ALS Cognitive Behavioral Screen (ALS-CBS) and Frontal Assessment Battery (FAB) between the probiotic and placebo groups over the 24 weeks of intervention.
Change in FAB score | 24 weeks
  To compare the average change from baseline in ALS Cognitive Behavioral Screen (ALS-CBS) and Frontal Assessment Battery (FAB) between the probiotic and placebo groups over the 24 weeks of intervention.
Change in neurofilament light chain concentration | 24 weeks
  To compare the average change from baseline in the neurofilament light chain concentration between the probiotic and placebo groups over the 24 weeks of intervention.
Change in ALSAQ-5 scores | 24 weeks
  To compare the average change from baseline in the Amyotrophic Lateral Sclerosis Assessment Questionnaire-5 (ALSAQ-5) between the probiotic and placebo groups over the 24 weeks of intervention.
Change in fecal microbiota in ALS-FTDSD patients | 24 weeks
  To compare the fecal microbiota composition, diversity, and strain recovery over the 24 weeks of intervention in the probiotic and placebo groups. Techniques will be based on the extraction of DNA and amplification of 16S ribosomal RNA genes. These genes are highly conserved between bacterial species, but vary in a manner that allows species identification.
Polar metabolite profiles of healthy participants | 24 weeks
  To explore polar metabolite profiles from baseline in healthy participants over the 24 weeks of intervention. Targets will be key microbiota metabolites: trimethylamine N-oxide (TMAO), short-chain fatty acids, and metabolites derived from tryptophan.
Lipidomic profiles of healthy participants | 24 weeks
  To explore lipidomic profiles from baseline in healthy participants over the 24 weeks of intervention. This will be a lipid profiling and quantification by using mass-spectrometry-based lipidomics. We are going to test 900 different lipids, which can be classified in 20 classes ans subclasses of interest.
Fecal microbiota of healthy participants | 24 weeks
  Explore the fecal microbiota composition, diversity, and strain recovery over the 24 weeks in the healthy participants. Techniques will be based on the extraction of DNA and amplification of 16S ribosomal RNA genes. These genes are highly conserved between bacterial species, but vary in a manner that allows species identification.

OTHER OUTCOMES:
Number of AEs and SAEs | 28 weeks
  To compare the number of adverse events (AEs) and serious adverse events (SAEs) that occur among to the probiotic group versus the placebo group throughout the study.
Changes in lab safety marker: Complete Blood Count (CBC) | 24 weeks
  Changes (outside normal variation) in safety lab marker: Complete Blood Count (CBC).
Changes in lab safety markers: Liver Function Test (LFT) - ALT | 24 weeks
  Changes (outside normal variation) in safety lab markers :Liver Function Tests (LFTs), more precisely alanine transaminase (ALT).
Changes in lab safety markers: Liver Function Test (LFT) - AST | 24 weeks
  Changes (outside normal variation) in safety lab markers :Liver Function Tests (LFTs), more precisely aspartate transaminase (AST).
Changes in lab safety markers: Liver Function Test (LFT) - bilirubin | 24 weeks
  Changes (outside normal variation) in safety lab markers :Liver Function Tests (LFTs), more precisely total bilirubin.
Changes in lab safety marker: creatinine | 24 weeks
  Changes (outside normal variation) in safety lab marker: creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Matte, MDCM, FRCP, Principal Investigator — CRCHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No